CLINICAL TRIAL: NCT02943811
Title: Effect of Uterine Manipulator on Recurrence and Mortality of Endometrial Cancer: a Multi-centric Study
Brief Title: Effect of Uterine Manipulator on Recurrence and Mortality of Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Doctor, Università degli Studi dell'Insubria
Other Study IDs: 521
Record Dates: First submitted 2016-10-22; First posted 2016-10-25 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; survival; uterine manipulator
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MANIPULATOR: Patients who were operated for endometrial cancer by laparoscopy with the use of a uterine manipulator
  Interventions: Device: UTERINE MANIPULATOR
- NO MANIPULATOR: Patients who were operated for endometrial cancer by laparoscopy without the use of a uterine manipulator

INTERVENTIONS:
Device: UTERINE MANIPULATOR — Patients were operated laparoscopically with the aid or not of an intrauterine probe to manipulate the uterus
  Groups: MANIPULATOR

SUMMARY:
The investigators sought to retrospectively assess whether the use of a intrauterine device to manipulate the uterus does affect the long-term oncologic outcomes of patients operated by laparoscopy for endometrial cancer

DETAILED DESCRIPTION:
The investigators retrospectively collected data regarding patients who received operation by laparoscopy for presumed clinical stage I endometrial cancer. The subjects were then stratified according to the use or not of the uterine manipulator. The investigators also considered the actual type of manipulator used. Then disease-free, disease-specific and overall survival were evaluated, as well as all the possible factors associated with prognosis.

Data were retrieved from specifically designed research quality internal surgical databases, prospectively updated by trained residents on a regular basis, in order to capture all the possible surgical and follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage I endometrial cancer
* Laparoscopic operation

Exclusion Criteria:

* post-operative oncologic follow-up < 12 months
* extra-uterine evidence of disease

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women affected by early endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 951 (Actual)
Dates: Start 2016-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Disease recurrence | 4 years
  Relapse of disease during follow-up

SECONDARY OUTCOMES:
disease specific survival | 4 years
  Kaplan Meyer curves and Log-rank test to explore disease-specific survival
overall survival | 4 years
  Kaplan Meyer curves and Log-rank test to explore overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, Principal Investigator — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcos-Sanmartin J, Lopez Fernandez JA, Sanchez-Paya J, Pinero-Sanchez OC, Roman-Sanchez MJ, Quijada-Cazorla MA, Candela-Hidalgo MA, Martinez-Escoriza JC. Does the Type of Surgical Approach and the Use of Uterine Manipulators Influence the Disease-Free Survival and Recurrence Rates in Early-Stage Endometrial Cancer? Int J Gynecol Cancer. 2016 Nov;26(9):1722-1726. doi: 10.1097/IGC.0000000000000808. PMID 27518143
- [Background] Tinelli R, Cicinelli E, Tinelli A, Bettocchi S, Angioni S, Litta P. Laparoscopic treatment of early-stage endometrial cancer with and without uterine manipulator: Our experience and review of literature. Surg Oncol. 2016 Jun;25(2):98-103. doi: 10.1016/j.suronc.2016.03.005. Epub 2016 Mar 23. PMID 27312035